CLINICAL TRIAL: NCT05096156
Title: Evaluation of Wear Experience With PRECISION1® Contact Lenses in Biofinity® Contact Lens Wearers
Brief Title: Evaluation of Wear Experience With Daily Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, PI, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021H0118
Record Dates: First submitted 2021-10-19; First posted 2021-10-27 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Contact Lens

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All participants are fit with the study daily disposable lenses (Experimental): All subjects are re-fit into their habitual monthly replacement contact lenses. Subjects are requested to wear the lenses for one week, for a minimum of at least 6 hours per day for 5 days. Upon return, subjects are refit into the daily disposable contact lenses.
  Interventions: Device: Precision1® Daily Disposable Contact Lens

INTERVENTIONS:
Device: Precision1® Daily Disposable Contact Lens — Soft, spherical contact lens used to correct distance vision.

SUMMARY:
To evaluate the wear experience of current monthly replacement contact lens wearers after they have been fit into a daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Currently wear Biofinity® monthly replacement spherical contact lenses.
* Distance visual acuity of 20/25 or better with current contact lenses.
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI).
* Ability to give informed consent.
* Willing to spend time for the study, which includes attending two study visits and wearing contact lenses on days between study visits.

Exclusion Criteria:

* No current ocular inflammation or infection.
* Not currently pregnant or lactating.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants Are Fit With the Study Daily Disposable Lenses
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants Are Fit With the Study Daily Disposable Lenses
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Subjective Assessment of Precision1® Daily Disposable Contact Lens
Description: Contact Lens Dry Eye Questionnaire (CLDEQ) survey (0-37, with higher scores related to higher symptoms)
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | All Participants Are Fit With the Study Daily Disposable Lenses
Number analyzed (Participants) | 30
units on a scale | 6.5 [3 to 10]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- All Participants: All subjects are re-fit into their habitual monthly replacement contact lenses. Subjects are requested to wear the lenses for one week, for a minimum of at least 6 hours per day for 5 days. Upon return, subjects are refit into the Verofilcon A daily disposable study contact lenses.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT05096156/Prot_SAP_002.pdf